CLINICAL TRIAL: NCT00000552
Title: Shock Trial: Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 96; R01HL049970 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia; Shock, Cardiogenic
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia; Shock, Cardiogenic | interventions — Angioplasty, Balloon, Coronary; Coronary Artery Bypass; Thrombolytic Therapy

INTERVENTIONS:
Procedure: angioplasty, transluminal, percutaneous coronary
Procedure: coronary artery bypass
Drug: thrombolytic therapy

SUMMARY:
To test if early revascularization, primarily with angioplasty (PTCA) or bypass surgery (CABG), reduced all-cause in-hospital mortality from cardiogenic shock compared to conventional treatment, including thrombolysis.

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 7.5 percent of all acute myocardial infarctions which are diagnosed in an emergency room or in-hospital lead to cardiogenic shock and an in-hospital death rate of 70 to 80 percent, usually within one to two days of diagnosis of cardiogenic shock. The high death rate has not changed in the last two decades. Non-random clinical series and animal studies suggest that rapid revascularization following cardiogenic shock complicating acute myocardial infarction may substantially improve survival. However, the apparent benefit reported in the non-random clinic studies could have resulted partly from a selection bias towards patients with a better prognosis.

DESIGN NARRATIVE:

Randomized, multicenter, Phase III, controlled clinical trial. Patients with shock due to left ventricular failure complicating myocardial infarction were randomly assigned to emergency revascularization or initial medical stabilization. Revascularization was accomplished by either coronary-artery bypass grafting or angioplasty. A total of 152 patients were randomized to early revascularization and 150 patients to conventional therapy consisting of thrombolytics and a possible late attempt at revascularization. Intraaortic balloon counterpulsation was performed in 86 percent of the patients in both groups. The primary endpoint was mortality from all causes at 30 days. Secondary endpoints included all-cause mortality at six months and assessment of the quality of life in survivors after discharge.

All patients with a clinically suspected diagnosis of cardiogenic shock complicating myocardial infarction formed a registry, with limited information collected on in-hospital procedures, medications, length of stay and vital status at discharge.

The study has been extended through June, 2005 for patient follow-up and data analyses. Long-term survival rates (6 to 11 years post-MI) will be estimated and the quality of life of survivors of acute MI complicated by cardiogenic shock will be studied. Extended trial data analyses will be conducted: a) To determine the early echocardiographic parameters which are associated with one year survival in cardiogenic shock patients, and to assess the interaction of these parameters with early revascularization; b) To examine differences in disease course and patient outcome as a function of age, gender, national practice, and changes in serial hemodynamic measurements, as well as to better characterize the related conditions and complications of cardiogenic shock.

ELIGIBILITY:
Men and women with myocardial infarction and cardiogenic shock.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sleeper — New England Research Institute, Inc.

REFERENCES:
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Ryan TJ. Early revascularization in cardiogenic shock--a positive view of a negative trial. N Engl J Med. 1999 Aug 26;341(9):687-8. doi: 10.1056/NEJM199908263410910. No abstract available. PMID 10460822
- [Background] Menon V, Webb JG, Hillis LD, Sleeper LA, Abboud R, Dzavik V, Slater JN, Forman R, Monrad ES, Talley JD, Hochman JS. Outcome and profile of ventricular septal rupture with cardiogenic shock after myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries in cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1110-6. doi: 10.1016/s0735-1097(00)00878-0. PMID 10985713
- [Background] Thompson CR, Buller CE, Sleeper LA, Antonelli TA, Webb JG, Jaber WA, Abel JG, Hochman JS. Cardiogenic shock due to acute severe mitral regurgitation complicating acute myocardial infarction: a report from the SHOCK Trial Registry. SHould we use emergently revascularize Occluded Coronaries in cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1104-9. doi: 10.1016/s0735-1097(00)00846-9. PMID 10985712
- [Background] Shindler DM, Palmeri ST, Antonelli TA, Sleeper LA, Boland J, Cocke TP, Hochman JS. Diabetes mellitus in cardiogenic shock complicating acute myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1097-103. doi: 10.1016/s0735-1097(00)00877-9. PMID 10985711
- [Background] Jacobs AK, French JK, Col J, Sleeper LA, Slater JN, Carnendran L, Boland J, Jiang X, LeJemtel T, Hochman JS. Cardiogenic shock with non-ST-segment elevation myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded coronaries for Cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1091-6. doi: 10.1016/s0735-1097(00)00888-3. PMID 10985710
- [Background] Hochman JS, Sleeper LA, Godfrey E, McKinlay SM, Sanborn T, Col J, LeJemtel T. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK: an international randomized trial of emergency PTCA/CABG-trial design. The SHOCK Trial Study Group. Am Heart J. 1999 Feb;137(2):313-21. doi: 10.1053/hj.1999.v137.95352. PMID 9924166
- [Background] Wong SC, Sanborn T, Sleeper LA, Webb JG, Pilchik R, Hart D, Mejnartowicz S, Antonelli TA, Lange R, French JK, Bergman G, LeJemtel T, Hochman JS. Angiographic findings and clinical correlates in patients with cardiogenic shock complicating acute myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1077-83. doi: 10.1016/s0735-1097(00)00873-1. PMID 10985708
- [Background] Webb JG, Sleeper LA, Buller CE, Boland J, Palazzo A, Buller E, White HD, Hochman JS. Implications of the timing of onset of cardiogenic shock after acute myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1084-90. doi: 10.1016/s0735-1097(00)00876-7. PMID 10985709
- [Background] Slater J, Brown RJ, Antonelli TA, Menon V, Boland J, Col J, Dzavik V, Greenberg M, Menegus M, Connery C, Hochman JS. Cardiogenic shock due to cardiac free-wall rupture or tamponade after acute myocardial infarction: a report from the SHOCK Trial Registry. Should we emergently revascularize occluded coronaries for cardiogenic shock? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1117-22. doi: 10.1016/s0735-1097(00)00845-7. PMID 10985714
- [Background] Menon V, White H, LeJemtel T, Webb JG, Sleeper LA, Hochman JS. The clinical profile of patients with suspected cardiogenic shock due to predominant left ventricular failure: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries in cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1071-6. doi: 10.1016/s0735-1097(00)00874-3. PMID 10985707
- [Background] Menon V, Slater JN, White HD, Sleeper LA, Cocke T, Hochman JS. Acute myocardial infarction complicated by systemic hypoperfusion without hypotension: report of the SHOCK trial registry. Am J Med. 2000 Apr 1;108(5):374-80. doi: 10.1016/s0002-9343(00)00310-7. PMID 10759093
- [Background] Hochman JS, Buller CE, Sleeper LA, Boland J, Dzavik V, Sanborn TA, Godfrey E, White HD, Lim J, LeJemtel T. Cardiogenic shock complicating acute myocardial infarction--etiologies, management and outcome: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1063-70. doi: 10.1016/s0735-1097(00)00879-2. PMID 10985706
- [Background] Sanborn TA, Sleeper LA, Bates ER, Jacobs AK, Boland J, French JK, Dens J, Dzavik V, Palmeri ST, Webb JG, Goldberger M, Hochman JS. Impact of thrombolysis, intra-aortic balloon pump counterpulsation, and their combination in cardiogenic shock complicating acute myocardial infarction: a report from the SHOCK Trial Registry. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? J Am Coll Cardiol. 2000 Sep;36(3 Suppl A):1123-9. doi: 10.1016/s0735-1097(00)00875-5. PMID 10985715
- [Background] Hochman JS, Sleeper LA, White HD, Dzavik V, Wong SC, Menon V, Webb JG, Steingart R, Picard MH, Menegus MA, Boland J, Sanborn T, Buller CE, Modur S, Forman R, Desvigne-Nickens P, Jacobs AK, Slater JN, LeJemtel TH; SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. One-year survival following early revascularization for cardiogenic shock. JAMA. 2001 Jan 10;285(2):190-2. doi: 10.1001/jama.285.2.190. PMID 11176812
- [Background] Webb JG, Sanborn TA, Sleeper LA, Carere RG, Buller CE, Slater JN, Baran KW, Koller PT, Talley JD, Porway M, Hochman JS; SHOCK Investigators. Percutaneous coronary intervention for cardiogenic shock in the SHOCK Trial Registry. Am Heart J. 2001 Jun;141(6):964-70. doi: 10.1067/mhj.2001.115294. PMID 11376311
- [Background] Carnendran L, Abboud R, Sleeper LA, Gurunathan R, Webb JG, Menon V, Dzavik V, Cocke T, Hochman JS. Trends in cardiogenic shock: report from the SHOCK Study. The SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK? Eur Heart J. 2001 Mar;22(6):472-8. doi: 10.1053/euhj.2000.2312. PMID 11237542
- [Background] Wong SC, Sleeper LA, Monrad ES, Menegus MA, Palazzo A, Dzavik V, Jacobs A, Jiang X, Hochman JS; SHOCK Investigators. Absence of gender differences in clinical outcomes in patients with cardiogenic shock complicating acute myocardial infarction. A report from the SHOCK Trial Registry. J Am Coll Cardiol. 2001 Nov 1;38(5):1395-401. doi: 10.1016/s0735-1097(01)01581-9. PMID 11691514
- [Background] Menon V, Fincke R. Cardiogenic shock: a summary of the randomized SHOCK trial. Congest Heart Fail. 2003 Jan-Feb;9(1):35-9. doi: 10.1111/j.1751-7133.2003.tb00020.x. PMID 12556676
- [Background] Jacobs AK, Leopold JA, Bates E, Mendes LA, Sleeper LA, White H, Davidoff R, Boland J, Modur S, Forman R, Hochman JS. Cardiogenic shock caused by right ventricular infarction: a report from the SHOCK registry. J Am Coll Cardiol. 2003 Apr 16;41(8):1273-9. doi: 10.1016/s0735-1097(03)00120-7. PMID 12706920
- [Background] Picard MH, Davidoff R, Sleeper LA, Mendes LA, Thompson CR, Dzavik V, Steingart R, Gin K, White HD, Hochman JS; SHOCK Trial. SHould we emergently revascularize Occluded Coronaries for cardiogenic shocK. Echocardiographic predictors of survival and response to early revascularization in cardiogenic shock. Circulation. 2003 Jan 21;107(2):279-84. doi: 10.1161/01.cir.0000045667.11911.f6. PMID 12538428
- [Background] Dzavik V, Sleeper LA, Cocke TP, Moscucci M, Saucedo J, Hosat S, Jiang X, Slater J, LeJemtel T, Hochman JS; SHOCK Investigators. Early revascularization is associated with improved survival in elderly patients with acute myocardial infarction complicated by cardiogenic shock: a report from the SHOCK Trial Registry. Eur Heart J. 2003 May;24(9):828-37. doi: 10.1016/s0195-668x(02)00844-8. PMID 12727150
- [Background] Webb JG, Lowe AM, Sanborn TA, White HD, Sleeper LA, Carere RG, Buller CE, Wong SC, Boland J, Dzavik V, Porway M, Pate G, Bergman G, Hochman JS; SHOCK Investigators. Percutaneous coronary intervention for cardiogenic shock in the SHOCK trial. J Am Coll Cardiol. 2003 Oct 15;42(8):1380-6. doi: 10.1016/s0735-1097(03)01050-7. PMID 14563578
- [Background] Sanborn TA, Sleeper LA, Webb JG, French JK, Bergman G, Parikh M, Wong SC, Boland J, Pfisterer M, Slater JN, Sharma S, Hochman JS; SHOCK Investigators. Correlates of one-year survival inpatients with cardiogenic shock complicating acute myocardial infarction: angiographic findings from the SHOCK trial. J Am Coll Cardiol. 2003 Oct 15;42(8):1373-9. doi: 10.1016/s0735-1097(03)01051-9. PMID 14563577
- [Background] French JK, Feldman HA, Assmann SF, Sanborn T, Palmeri ST, Miller D, Boland J, Buller CE, Steingart R, Sleeper LA, Hochman JS; SHOCK Investigators. Influence of thrombolytic therapy, with or without intra-aortic balloon counterpulsation, on 12-month survival in the SHOCK trial. Am Heart J. 2003 Nov;146(5):804-10. doi: 10.1016/S0002-8703(03)00392-2. PMID 14597928
- [Background] Fincke R, Hochman JS, Lowe AM, Menon V, Slater JN, Webb JG, LeJemtel TH, Cotter G; SHOCK Investigators. Cardiac power is the strongest hemodynamic correlate of mortality in cardiogenic shock: a report from the SHOCK trial registry. J Am Coll Cardiol. 2004 Jul 21;44(2):340-8. doi: 10.1016/j.jacc.2004.03.060. PMID 15261929
- [Background] White HD, Palmeri ST, Sleeper LA, French JK, Wong CK, Lowe AM, Crapo JW, Koller PT, Baran KW, Boland JL, Hochman JS, Wagner GS; SHOCK Trial Investigators. Electrocardiographic findings in cardiogenic shock, risk prediction, and the effects of emergency revascularization: results from the SHOCK trial. Am Heart J. 2004 Nov;148(5):810-7. doi: 10.1016/j.ahj.2004.05.012. PMID 15523311
- [Background] Sleeper LA, Ramanathan K, Picard MH, Lejemtel TH, White HD, Dzavik V, Tormey D, Avis NE, Hochman JS; SHOCK Investigators. Functional status and quality of life after emergency revascularization for cardiogenic shock complicating acute myocardial infarction. J Am Coll Cardiol. 2005 Jul 19;46(2):266-73. doi: 10.1016/j.jacc.2005.01.061. PMID 16022953
- [Background] Kohsaka S, Menon V, Lowe AM, Lange M, Dzavik V, Sleeper LA, Hochman JS; SHOCK Investigators. Systemic inflammatory response syndrome after acute myocardial infarction complicated by cardiogenic shock. Arch Intern Med. 2005 Jul 25;165(14):1643-50. doi: 10.1001/archinte.165.14.1643. PMID 16043684
- [Background] White HD, Assmann SF, Sanborn TA, Jacobs AK, Webb JG, Sleeper LA, Wong CK, Stewart JT, Aylward PE, Wong SC, Hochman JS. Comparison of percutaneous coronary intervention and coronary artery bypass grafting after acute myocardial infarction complicated by cardiogenic shock: results from the Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock (SHOCK) trial. Circulation. 2005 Sep 27;112(13):1992-2001. doi: 10.1161/CIRCULATIONAHA.105.540948. PMID 16186436
- [Background] Palmeri ST, Lowe AM, Sleeper LA, Saucedo JF, Desvigne-Nickens P, Hochman JS; SHOCK Investigators. Racial and ethnic differences in the treatment and outcome of cardiogenic shock following acute myocardial infarction. Am J Cardiol. 2005 Oct 15;96(8):1042-9. doi: 10.1016/j.amjcard.2005.06.033. Epub 2005 Aug 22. PMID 16214435
- [Background] Dzavik V, Sleeper LA, Picard MH, Sanborn TA, Lowe AM, Gin K, Saucedo J, Webb JG, Menon V, Slater JN, Hochman JS; SHould we emergently revascularize Occluded Coronaries in cardiogenic shocK Investigators. Outcome of patients aged >or=75 years in the SHould we emergently revascularize Occluded Coronaries in cardiogenic shocK (SHOCK) trial: do elderly patients with acute myocardial infarction complicated by cardiogenic shock respond differently to emergent revascularization? Am Heart J. 2005 Jun;149(6):1128-34. doi: 10.1016/j.ahj.2005.03.045. PMID 15976798
- [Derived] Sleeper LA, Reynolds HR, White HD, Webb JG, Dzavik V, Hochman JS. A severity scoring system for risk assessment of patients with cardiogenic shock: a report from the SHOCK Trial and Registry. Am Heart J. 2010 Sep;160(3):443-50. doi: 10.1016/j.ahj.2010.06.024. PMID 20826251
- [Derived] Hochman JS, Sleeper LA, Webb JG, Dzavik V, Buller CE, Aylward P, Col J, White HD; SHOCK Investigators. Early revascularization and long-term survival in cardiogenic shock complicating acute myocardial infarction. JAMA. 2006 Jun 7;295(21):2511-5. doi: 10.1001/jama.295.21.2511. PMID 16757723